CLINICAL TRIAL: NCT00904332
Title: Changes in the Posterior Parietal Cortex - Primary Motor Cortex Pathway Induced by Motor Training
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090146; 09-N-0146
Record Dates: First submitted 2009-05-16; First posted 2009-05-19 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-12-29

CONDITIONS: Movement Disorders; Heathly Subjects
Keywords: Transcranial Magnetic Stimulation (TMS); Electroencephalogram (EEG); Motor Learning; Health Volunteer; HV
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Objective

When learning to tap to a rhythm the brain has to coordinate information from different senses (eyes, ears, touch). This information has to be integrated into a movement plan to allow a smooth, continuous performance. Two brain areas that are of particular interest for this task are the posterior parietal cortex that integrates sensory and motor information and the primary motor cortex that sends out the movement commands to the muscles. These areas communicate via nerve connections with each other. The goal of this research proposal is to examine if the strength of the connection between those areas can be changed by practicing a simple tapping task and if the change in connection strength depends on if the rhythms were shown by visual or auditory stimuli. Additionally we will investigate how the ability to tap rhythms relates to other cognitive abilities like problem solving.

Study Population

We intend to study 20 adult healthy volunteers on an outpatient basis.

Design

In three experimental sessions we propose to use transcranial magnetic stimulation (TMS) and electro encephalography (EEG) to examine the role of the posterior parietal cortex in motor learning. In session 1 a neurological examination will be performed and a clinical and anatomical MRI (Magnet Resonance Image) will be taken. Session 1 can be skipped if an MRI and a neurological exam have been performed at the NIH during the last year. In session 2 TMS will be used to examine the connection between posterior parietal cortex and primary motor cortex before and after rhythm training. Additionally, EEG will be recorded during the training session. In session 3 we will examine how the ability to tap to different beats relates to higher cognitive functions. We will record EEG during tapping simple beats and we will administer a pen and paper problem-solving test.

Outcome Measures

In session 2 the primary outcome measure will be change in conditioned Motor Evoked Potential (MEP) peak-to-peak amplitude after learning temporal motor sequences measured in the primary motor cortex. A secondary outcome measure will be the interregional coherence changes as measured by EEG during training. In session 3 the primary outcome will be performance on the tapping task and on the pen and paper test as well as the interregional coherence changes as measured by EEG during the tapping task.

DETAILED DESCRIPTION:
Objective

When learning to tap to a rhythm the brain has to coordinate information from different senses (eyes, ears, touch). This information has to be integrated into a movement plan to allow a smooth, continuous performance. Two brain areas that are of particular interest for this task are the posterior parietal cortex that integrates sensory and motor information and the primary motor cortex that sends out the movement commands to the muscles. These areas communicate via nerve connections with each other. The goal of this research proposal is to examine if the strength of the connection between those areas can be changed by practicing a simple tapping task and if the change in connection strength depends on if the rhythms were shown by visual or auditory stimuli. Additionally we will investigate how the ability to tap rhythms relates to other cognitive abilities like problem solving.

Study Population

We intend to study 20 adult healthy volunteers on an outpatient basis.

Design

In three experimental sessions we propose to use transcranial magnetic stimulation (TMS) and electro encephalography (EEG) to examine the role of the posterior parietal cortex in motor learning. In session 1 a neurological examination will be performed and a clinical and anatomical MRI (Magnet Resonance Image) will be taken. Session 1 can be skipped if an MRI and a neurological exam have been performed at the NIH during the last year. In session 2 TMS will be used to examine the connection between posterior parietal cortex and primary motor cortex before and after rhythm training. Additionally, EEG will be recorded during the training session. In session 3 we will examine how the ability to tap to different beats relates to higher cognitive functions. We will record EEG during tapping simple beats and we will administer a pen and paper problem-solving test.

Outcome Measures

In session 2 the primary outcome measure will be change in conditioned Motor Evoked Potential (MEP) peak-to-peak amplitude after learning temporal motor sequences measured in the primary motor cortex. A secondary outcome measure will be the interregional coherence changes as measured by EEG during training. In session 3 the primary outcome will be performance on the tapping task and on the pen and paper test as well as the interregional coherence changes as measured by EEG during the tapping task.

ELIGIBILITY:
* INCLUSION:
* Age over 18 years
* Absence of any neurologic condition that might affect performance of the tasks in these experiments
* Right handedness

EXCLUSION:

* Taking medications which include antidepressants, anxiolytics, anticonvulsants, antipsychotics, antiparkinson, hypnotics, stimulants, and/or antihistamines
* Received botulinum toxin injection within 3 months of starting the protocol
* History of seizure disorder
* Presence of implanted devised such as pacemakers, medication pumps or defibrillators, metal in the cranium except mouth, intracardiac lines, history of shrapnel injury or any other condition/device that may contraindicated or prevent the acquisition of MRI
* A serious medical illness which prevents them from lying flat for up to 60 minutes
* Claustrophobia (fear of tight spaces), which prevents them from lying still in a tight or small space for up to 40 minutes
* Five years or more of formal musical education in any instrument
* Current pregnancy
* Known hearing loss

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-05-14; Study Completion 2011-12-29

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Andrew C, Pfurtscheller G. Event-related coherence as a tool for studying dynamic interaction of brain regions. Electroencephalogr Clin Neurophysiol. 1996 Feb;98(2):144-8. doi: 10.1016/0013-4694(95)00228-6. PMID 8598174
- [Background] Andrew C, Pfurtscheller G. Dependence of coherence measurements on EEG derivation type. Med Biol Eng Comput. 1996 May;34(3):232-8. doi: 10.1007/BF02520079. PMID 8762831
- [Background] Baumer T, Bock F, Koch G, Lange R, Rothwell JC, Siebner HR, Munchau A. Magnetic stimulation of human premotor or motor cortex produces interhemispheric facilitation through distinct pathways. J Physiol. 2006 May 1;572(Pt 3):857-68. doi: 10.1113/jphysiol.2006.104901. PMID 16497712